CLINICAL TRIAL: NCT06527443
Title: Arterial Stiffness as a Predictor of Acute Kidney Injury in Patients With Sepsis
Brief Title: Arterial Stiffness in Patients With Sepsis
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Ali Ahmed, assistant professor of internal medicine, Assiut University
Other Study IDs: AssiutU sepsis
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: the Arterial Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute kidney injury
- non acute kidney injury

SUMMARY:
To investigate whether arterial stiffness, as defined by measuring Pulse Wave Velocity, could be identified as an independent risk factor for development of acute kidney injury in sepsis.

To compare between the Pulse Wave Velocity and shear wave ultrasound elastography (SWE) as a different methods of evaluation of arterial stiffness in prediction of acute kidney injury in sepsis.

DETAILED DESCRIPTION:
Demographic and historical data: the patient age, sex, history of hypertension, diabetes ,peripheral vascular disease , IHD, source of sepsis and indication of mechanical ventilation if indicated.

Clinical examination data: pulse, blood pressure, respiratory rate, temperature and thorough chest, cardiac and neurological examination data will be obtained.

Volume state of the patient: CVP measurement, input and output fluid chart. Investigation : CBC( Neutrophil count, Neutrophil/lymphocyte ratio), Blood urea and serum creatinine ,serum electrolytes, serum lactate,serum albumin,CRP ,coagualtion profile and lipid profile. sequential organ failure assessment (SOFA) score, acute physiology and chronic health evaluation (APACHE II) score, and complete sepsis workup to identify the possible sources of sepsis.

12 lead ECG and Echocardiographic data that include: Left and right atrial dimensions. The left ventricular ejection fraction will be assessed by the Simpson method, left ventricular diastolic function will be assessed by measuring velocities of the mitral E and A waves and of the e' wave of the external mitral annulus and by calculating the E/e' ratio. Right ventricle dimension and dysfunction will be evaluated by TAPSE and pulmonary artery acceleration time. Pulmonary artery pressure will be measured from Tricuspid flow if possible.

Pulse Wave Velocity (PWV), a measurement of arterial stiffness, will be assessed at the systemic region (carotid-femoral PWV), which is the gold standard method. In the first 24 hours of admission.

The two-dimensional SWE technique will be used in our study , an imaging method will be obtained by simultaneously applying multiple ARFI waves into the tissue and measuring the resulting shear waves .It will be assessed in the first 24 hours of admission.

RRI will be measured at the time of admission. All measurements will be performed by the same examiner and repeated by an independent blinded operator. Using pulse-wave Doppler, an interlobar or arcuate artery will be selected. RRI will be calculated as the equation "(PSV-EDV)/PSV". The means of three distinct RRI calculations will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who admitted to critical care unit of Internal medicine department with sepsis after obtaining consent.

Exclusion Criteria:

* Children below 18 yr.
* Patients could not be scanned within 24-h after ICU admission.
* Patients with end stage renal disease or transplanted kidney.
* patients with renal artery stenosis, and obstructive uropathy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who admitted to critical care unit of Internal medicine department with sepsis after obtaining consent. Demographic data Clinical examination data will be obtained.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness in prediction of AKI in patients with sepsis | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dina Ali Hamad, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No